CLINICAL TRIAL: NCT04240873
Title: Randomized Double-blind Clinical Study of Intra Articular Injection of Catholic MASTER Cell in Knee Osteoarthritis
Brief Title: Clinical Study of Intra Articular Injection of Catholic MASTER Cell (Bone Marrow Derived Mesenchymal Stem Cell) in Knee Osteoarthritis
Acronym: MSC-OA
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul St. Mary's Hospital (Other)
Responsible Party: Principal Investigator, Ji Hyeon Ju, Professor, Seoul St. Mary's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KC19CNSI0469
Record Dates: First submitted 2019-12-10; First posted 2020-01-27 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Osteoarthritis, Knee
Keywords: osteoarthritis; mesenchymal stem cell
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MASTER cell (Experimental): Intraarticular injection of Catholic MASTER cell, 1 time, 1 x 10^8 cells/DMEM 5cc, into knee joint of patients with osteoarthritis
  Interventions: Biological: Catholic MASTER cell
- Saline (Placebo Comparator): Intraarticular injection of saline, 1 time, 5cc, into knee joint of patients with osteoarthritis
  Interventions: Other: Saline

INTERVENTIONS:
Biological: Catholic MASTER cell — Injection of CATHOLIC MASTER cells 1 x 10^8 cells/DMEM 5cc into knee of patents with osteoarthritis
  Arms: MASTER cell
Other: Saline — Injection of saline 5cc into knee of patents with osteoarthritis
  Arms: Saline

SUMMARY:
1. objective

   - safety and efficacy evalaution of MASTER cells injected into knee of patients with osteoarthritis
2. background

   * osteoarthritis

     * Osteoarthritis is severe and intractable musculoskeletal disease that eventually leads to joint failure and pain due to inflammation and joint injury.
     * OA is one of the most prevalent diseases. The prevalence increases with age, but overuse and trauma can result in OA in young population as well.
     * Injured cartilage can not be regenerated spontaneously, untreated injured cartilage eventually leads to osteoarthritis. Surgical treatment may repair the damage but the reparied cartilage may turn out to be fibrocartilage rather than hyaline cartilage.
   * Curent treatment

     * medical therapy: medication for symptom relief, together with exercise. Medications include NSAIDS visco-supplement.
     * surgical therapy: total knee replacement arthroplasty
     * to overcome such limitations, cell therapy such as stem cell/ chondrocyte injection is being investigated
3. Hypothesis

   - Intra articular injection of MASTER cells will show safety and efficacy in terms of pain and functional improvement.
4. Protocol 1) deisgn : Injection of MASTER cell 1X 10^8 cells/2cc (experimental arm) or 2cc saline (placebo arm) into knee of patients with osteoarthritis 2) outcomes

   * primary outcome : safety evaluation(adverse event)
   * secondary outcomes : check on 1,2,3,6,9,12 months, atient reported outcome (WOMAC, KOOS, IKDC, pain VAS) 3,12 months SF-36, knee MRI score, serum cytokine, bone turnover marker 12 months x-ray 3) Disease
   * osteoarthritis

     4) Subjects
     1. inclusion : age 20-80yrs, diagnosed with OA according to ACR criteria for knee OA, baseline pain VAS equal or more than 50mm
     2. exclusion: lower extremities surgery within 6months or planned surgery, concommitant systemic rheumatic diseases that can affect the results of the trial, steroid intraarticular inejction into the index knee within 3months, clinicallly meaningful abnormal lab tests (liver function, kidney function)

     5) evaluation
   * primary outome : compare the number and proportion of of adverse event and lab test abnormalities between the two arms
   * secondary outome

     1. change of 100mm pain VAS
     2. change of Western Ontario and McMAster Universities Osteoarthritis (WOMAC) pain VAS, IKDC, KOOS total score
     3. change WOMAC sub scale, IKDC, KOOS
     4. chagne of KHAQ
     5. change of MRI indices
     6. change of x-ray( joins space narrowing)
     7. change of serum ESR/CRP, CTX-II

ELIGIBILITY:
Inclusion Criteria:

1. Age 20-80
2. diagnosed with knee osteoarthritis (OA) according to ACR classfication criteia for knee OA
3. symptomatic OA that lastede for at least 3 months before screening
4. Baseline Pain VAS ≥50 mm
5. treated with medication such as acetaminophen, tramadol, NSAID for at least 1month due to OA pain
6. X-ray Kellgren-Lawrence grade 1~4
7. volauntarily enrolled with informed consent
8. no improvement with medical treatment for at least 3 months

Exclusion Criteria:

1. disease in spine or lower extremities that can affect the outcome of index knee
2. surgery on lower extremities within 6month before injection or planned
3. joint symptoms that can affect the interpretation of the trial data or prevent the subject from enrollement including but not limited to symptomatic fracture, fibromyalgia, rheumatoid arthritis, reactive arthritis
4. steroid injection to the index knee within preivious 3months
5. hyaluronic acid injection to the index knee within preivious 6months
6. underwent cell therapy or gene therapy in the past
7. more than 3 times upper normal limit in one or more of the followings: serum creatinine, bilirubin, alanine aminotransferase (ALT) or aspartate aminotransferase (AST) or more than 3 times upper normal limit in two or more of the followings: bilirubin, alanine aminotransferase (ALT) or aspartate aminotransferase (AST)
8. participation in a different clinical trial other than this within 4 weeks after initiation of the current study
9. use (reccuent use or addiction) of substances that can affect pain sensation such as narcotics
10. females of childbearing age who do not consent to effective contraceptive methods during the study period
11. pregnant or lactating woman
12. malignancy
13. considered to be inappropriate for the trial by investigators

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2019-11-15 (Actual); Primary Completion 2021-03-31 (Estimated); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
adverse event according to CTCAE 5.0, clinically meaningful abnormalites in laboratory tests (blood) | Change from Baseline blood abnormalities at 12 month
Western Ontario and McMaster Universities Arthritis Index (WOMAC) score | Change from Baseline WOMAC score at 12 month
Knee injury and Osteoarthritis Outcome Score (KOOS) | Change from Baseline KOOS score at 12 month
International knee documentation committee (IKDC) | Change from Baseline IKDC score at 12 month
Cartilage damage evaluation through knee MRI | Change from Baseline cartilage morphology at 12 month
SF-36 questionnaire | Change from Baseline SF-36 score at 12 month
Serum inflammatory cytokine, acute phase reactant, bone turnover marker | Change from Baseline cytokine level, acute phase reactant, bone turnover marker level at 12 month
Cartilage damage evaluation through knee x-ray | Change from Baseline cartilage and bone morphology at 12 month

CONTACTS AND LOCATIONS:
Overall Officials: Ji Hyeon Ju, MD, PhD, Principal Investigator — The Catholic University of Korea
Locations (1):
- Catholic University of Korea, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided